CLINICAL TRIAL: NCT01211756
Title: Double-Blind, Randomized, Placebo-Controlled, Cross-Over Study of Intranasal Oxytocin Augmentation of Antidepressant Medication in Depressed Patients.
Brief Title: Oxytocin Add-on for Stable Depressed Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Break in funding
Sponsor: David Feifel (Other)
Responsible Party: Sponsor-Investigator, David Feifel, Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Oxytocin Depression
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2016-12

CONDITIONS: Major Depressive Disorder; Dysthymia Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Experimental): 20 IU of intranasal oxytocin twice per day for the first week, 40 IU of intranasal oxytocin twice per day for the following 3 weeks, one week wash out, 4 week placebo trial.
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Four week placebo trial, one week wash out, 20 IU of intranasal oxytocin twice per day for one week, 40 IU of intranasal oxytocin twice per day for 3 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — 20 IU BID for one week, followed by 40 IU BID for 3 weeks.
  Arms: Oxytocin
Drug: Placebo — 20 IU BID for one week, followed by 40 IU BID for 3 weeks.
  Arms: Placebo

SUMMARY:
The objective of the study is to compare the efficacy of intranasal oxytocin versus intranasal placebo to improve depression symptoms in patients with Major Depressive Disorder (MDD) or Dysthymia Disorder.

DETAILED DESCRIPTION:
Depression patients treated with even the best currently available antidepressant drugs continue to experience significant symptoms. There is a strong need for better treatments including treatments that can safely be given adjunctively with concurrent antidepressants in order to improve overall efficacy of treatment.

Oxytocin is a neurohypophyseal peptide best known for its role as a neurohormone involved in parturition and lactation. In addition to these well established peripheral effects, there is a compelling body of converging evidence indicating that oxytocin plays a critical role in the regulation of a number of diverse centrally-mediated behavioral and cognitive processes that are highly relevant to mood regulation and mood disorders, including social attachment (Argiolas and Gessa 1990; McCarthy and Aaltemus 1997).

Each subject will be enrolled for a 8 week treatment period after a screening phase. Study procedure involves weekly clinic visits as an outpatient. Twenty patients will be randomly assigned to either 40 IU oxytocin twice daily or vehicle placebo. After 4 weeks, treatments will be crossed over such that subjects that received oxytocin will receive placebo and vice versa. The study ratio is 1:1. Dose of oxytocin is based upon previous studies in humans showing improvement in psychiatric populations related changes in behavior and brain function (Kosfeld et al, 2005; Kirsch 2005; Heinrich M 2003).

The total study duration for each individual subject will be approximately 9 weeks, which includes up to 31-day screening period, a baseline (randomization) visit, four week treatment period, 1 week washout, baseline 2 visit, and four weeks cross over treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women, 18 years of age or older.
2. Meet DSM-IV criteria for Major Depressive Disorder or Dysthymia Disorder
3. Women of childbearing potential must test negative for pregnancy at the time of enrollment based on urine pregnancy test and agree to use a reliable method of birth control during the study.
4. Must be on a therapeutic dose of 1 or 2 antidepressants with no major dose changes for at least 4 weeks at randomization.
5. MADRS score of >17 at randomization
6. Have a Clinical Global Impressions-Severity (CGI-S) scale score of at least 4 (moderately ill) at baseline.
7. Must be able to communicate effectively with the investigator and study coordinator and have the ability to provide informed consent.
8. Must be able to use nasal spray
9. Must demonstrate an acceptable degree of compliance with medication and procedures in the opinion of the investigator. (If patient cannot then he/she will be considered for the acute only portion of this study.)

Permitted:

Subjects on up to 2 sleep medication (diphenhydramine, zolpidem, zaleplon, or diazepam), at a reasonable dose, as judged by the investigator, is permitted in this study.

Minor adjustments in sleep medication is acceptable. Patients will be asked to notify the study doctor of any changes to sleep aids.

Exclusion Criteria:

Subjects will be excluded from the study of they meet any of the following criteria:

1. Are pregnant or are breastfeeding (negative pregnancy test at screening)
2. A urine drug screen performed at screening must not show evidence of recent use of drugs of abuse
3. Any active medical condition that in the opinion of the investigator will interfere with the objectives of the study
4. Are unsuitable in any way to participate in this study, in the opinion of the investigator.
5. Another current DSM-IV diagnosis other than Major Depressive Disorder or Dysthymia Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-10; Primary Completion 2015-02 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Feifel, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: As there was only one subject enrolled, the results will not be analyzed.
Period: Overall Study
Arm/Group | All Participants
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The PI has left the institution and there was only one subject enrolled, the results will not be analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Total Score on Montgomery-Asberg Depression Rating Score (MADRS)
Description: The MADRS is a clinician-rated assessment used to measure the severity of depressive episodes in patients with mood disorders. The measure contains 10 items and each item is scored in a range of 0 to 6 points, with higher score indicating increased depressive symptoms.
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and there was only one subject enrolled, the results will not be analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Global Assessment of Functioning (GAF)
Description: The GAF considers psychological, social, and occupational functioning on a hypothetical continuum of mental health illness. Scores on the GAF range from 1 (extremely severe) to 100 (superior functioning).
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and there was only one subject enrolled, the results will not be analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Clinical Global Impression-Severity of Illness (CGI-S)
Description: The CGI-S is used to evaluate changes in overall severity of illness. Scores on the CGI-S range from 1 (not at all) to 7(among the most extremely ill).
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and there was only one subject enrolled, the results will not be analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Clinical Global Impression-Global Improvement (CGI-I)
Description: The CGI-I is a global assessment to evaluate the subjects' improvement or worsening from baseline. Scores on the CGI-I scale range from 1 (very much improved) to 7 (very much worse).
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and there was only one subject enrolled, the results will not be analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

5. Secondary Outcome: Young Mania Rating Scale (YMRS)
Description: The YMRS is an 11-item assessment used to assess the severity of mania in patients with a diagnosis of bipolar disorder. Ratings are based on patient self-reporting, combined with clinician observed.
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and there was only one subject enrolled, the results will not be analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: Hamilton-Anxiety Scale (HAM-A)
Description: The HAM-A is a clinician administered scale for the evaluation of anxiety symptoms. The HAM-A consists of 14 items of which each item is scored 0 (not present) to 4 (very severe).
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and there was only one subject enrolled, the results will not be analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

7. Secondary Outcome: Reading Trust in the Mind's Eye Test
Description: The subject will view approximately 16 faces and asked to rate trustfulness of the person in the picture.
Time Frame: Performed at the beginning and end of each treatment arm.
Population: The PI has left the institution and there was only one subject enrolled, the results will not be analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

8. Secondary Outcome: Profile of Mood States (POMS)
Description: The POMS is a self-rated scale to assess current mood states. The POMS consists of 65 words that the subject will rate from 1 (not at all) to 5 (extremely) based on how he/she feels at the time.
Time Frame: Performed at the beginning and end of each treatment arm
Population: The PI has left the institution and there was only one subject enrolled, the results will not be analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

9. Secondary Outcome: Arizona Sexual Experience Scale (ASEX)
Description: The ASEX is a self-rated scale to assess sexual functioning. The ASEX consists of 5 items that the subject will rate from 1 (Extremely strong, easily, or satisfying) to 6 (Absent or never) based on how he/she feels at the time.
Time Frame: Performed at each visit (weekly)
Population: The PI has left the institution and there was only one subject enrolled, the results will not be analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

10. Secondary Outcome: Peabody Picture Vocabulary Test
Description: The subject is read a series of words and is shown line drawings and is asked to match the word to the drawing.
Time Frame: Performed at the beginning of the study
Population: The PI has left the institution and there was only one subject enrolled, the results will not be analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

11. Secondary Outcome: California Verbal Learning Test
Description: The subject is read a list of words and asked to repeat them back first after the list is read and again 20 minutes later.
Time Frame: Performed at the beginning and end of each treatment arm
Population: The PI has left the institution and there was only one subject enrolled, the results will not be analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

12. Secondary Outcome: Letter Number Sequencing Memory Test
Description: The examinee is read a combination of numbers and letters and is asked to recall the numbers first in ascending order and then the letters in alphabetical order. Each item consists of three trials, and each trial is a different combination of numbers and letters.
Time Frame: Performed at the beginning and end of each treatment arm
Population: The PI has left the institution and there was only one subject enrolled, the results will not be analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

13. Secondary Outcome: Continuous Performance Test (CPT)
Description: Patients are told that they will see a series of letters presented on a screen. They are told to click a computer mouse only when they see the "target" stimulus, for instance the letter "X", and must refrain from clicking if they see any other letter presented.
Time Frame: Performed at the beginning and end of each treatment arm
Population: The PI has left the institution and there was only one subject enrolled, the results will not be analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The PI has left the institution and there was only one subject enrolled, the results will not be analyzed.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The PI has left the institution and there was only one subject enrolled, the results will not be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes